CLINICAL TRIAL: NCT02731287
Title: Efficacy and Safety of Topical Timolol Maleate 0.5% Solution for Superficial Infantile Hemangioma in Early Proliferative Phase. A Randomized Clinical Trial
Brief Title: Topical Timolol for Infantile Hemangioma in Early Proliferative Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-TIM-2013-156
Record Dates: First submitted 2015-11-17; First posted 2016-04-07 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Timolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Experimental): Timolol maleate 0.5% topical solution; 50% of the patients treated (randomized)
  Interventions: Drug: Timolol
- Placebo (Placebo Comparator): Saline topical solution; 50% of the patients treated (randomized)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Timolol — The patient will be treated with 2 drops twice a day over the lesion and rub with the finger (no occlusive) for 24 weeks
  Other Names: Timolol maleate 0.5%
  Arms: Timolol
Drug: Placebo — The patient will be treated with 2 drops twice a day over the lesion and rub with the finger (no occlusive) for 24 weeks
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
Infantile hemangioma (IH) is the most common benign vascular tumor in pediatric population. Oral propranolol is the treatment of choice for complicated hemangiomas. Topical timolol, a non-selective beta-blocker, is an emerging treatment which has been reported to be effective and safe for the treatment of IH, especially for superficial hemangiomas. Investigators hypothesize that treatment with topical timolol in the first two months of life, before the proliferative phase or in early proliferative phase, may prevent from further growing and the need to treat with oral propranolol.

DETAILED DESCRIPTION:
A multicentric, randomized, double-blind, placebo-controlled, phase II clinical trial to evaluate the efficacy and safety of 0.5% timolol maleate solution for the early treatment of infantile hemangioma.

Patients with less of 60 days of life with focal or segmental hemangiomas, superficial, mixed or abortive will be treated with topical timolol 0.5% twice a day for 24 weeks.

Changes in lesion size, color and thickness will be evaluated from photographs taken at 2,4,8,12,24 and 36 weeks. Vital signs and side effects will be recorded at each visit. Response to treatment will be evaluated by a blinded investigator in a semiquantitative scale (complete resolution, improve, stabilization, worsening).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for study participation and the use of the patient's photographs from the patient's parent(s) or guardian(s),
* The patient is between 10 and 60 days of age at the time of enrollment,
* The patient should have:

  * at least one focal or segmental hemangioma, mixed or superficial, present anywhere on the body of at least 0.3 cm of minimum diameter and not greater of 5 cm.
  * abortive or minimal growth hemangioma
  * Infantile hemangioma precursors

Exclusion Criteria:

* Patients > 60 days of age
* Complicated hemangiomas (life-threatening, function-threatening, or ulcerated)
* Children who have previously received systemic, intra-lesional or topical corticosteroids, imiquimod, vincristine, alpha-interferon, propranolol or other beta blockers, PDL laser.
* Patients with PHACES, LUMBAR, SACRAL or PELVIS syndrome.
* Internal involvement hemangiomas (liver, GI tract, larynx)
* Children with a personal history of asthma or cardiac conditions that may predispose to heart block.
* Children with congenital birth defects
* Children with Cancer (leukemia, sarcoma, neuroblastoma, retinoblastoma)
* Children with a history of hypersensitivity to beta blockers or excipients.

Ages: 10 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Complete or almost complete resolution of the lesions | 24 weeks
  Efficacy to treatment at 24 weeks, categorized as complete or almost complete resolution of the lesions (almost complete resolution defined as faint macular erythema, telangiectasia and no palpable component).
  This will be generated by independent blind evaluations by comparing photographs at baseline and 24 weeks. The investigators will score this improvement into one of the following categories (complete resolution, improve, stabilization, worsening)

SECONDARY OUTCOMES:
Adverse reactions | 24 weeks
  Evaluation of safety and adverse reactions. The investigators will monitor vital signs of the patients every follow-up visit and ask the caretakers about side effects and adverse reactions to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eulalia Baselga, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen del Rocío, Seville